CLINICAL TRIAL: NCT02726412
Title: Perioperative Mechanisms for Postoperative Function - Case of Lower Extremities Revascularisation
Brief Title: PACU Stay After Lower Limb Revascularisation
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Dr, DMSci, Rigshospitalet, Denmark
Other Study IDs: PACU revascularisation 2016
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Perioperative, Enhanced Recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Acute vs elective — non-intverention study

SUMMARY:
This study aims to describe the postoperative functions of patients with ischaemic lower extremities after undergoing revascularisation surgery . Primary endpoints will focus on complications in the post-anaesthesia care unit (PACU) which prevent discharge from PACU to the general ward. This include Aldrete scores and other complications that can be registrered descriptively. Furthermore, the study seeks to compare the complications outcomes between acute and elective revascularisation surgery.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of ischaemic lower extremities for instance intermittent claudication, resting leg pain, non-healing/gangrenouswounds and acute cold leg.
* Patients who underwent one or more of the following surgical procedure: PTA + TEA, TEA, bypass, thrombectomy, embolectomy, femoral-femoral crossover bypass, axillary-femoral bypass.

Exclusion Criteria:

* Only PTA intervention
* Only thrombolysis intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes every patients who undergo revascularisation surgery of one or both of lower extremeties to regain blood perfusion and relieve symptoms. The surgeries in question are for instance bypass, thrombectomy/embolectomy and thromboendarterectomy. The patients preoperative physical state for surgery will be registrered in detailed such as comorbidities, height, weight, bloodpressure and blood test results.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Complications assessed by aldrete score | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, abdominal center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided